CLINICAL TRIAL: NCT04202159
Title: PERPRISE: A Prospective Non-interventional Study Evaluating the Effectiveness of Perampanel (Fycompa®) as Only Add-on Treatment in Patients With Primary or Secondarily Generalized Tonic-clonic Seizures
Brief Title: A Study to Evaluate the Effectiveness of Perampanel as Only Add-on Treatment in Participants With Primary or Secondarily Generalized Tonic-clonic Seizures
Status: Completed | Type: Observational
Sponsor: Eisai GmbH (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M049-509
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Seizures
Keywords: E2007; Perampanel; Fycompa; Primary generalized tonic-clonic seizures; Secondarily generalized tonic-clonic seizures
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perampanel: Participants with PGTC or SGTC seizures may receive perampanel tablets or oral suspension as only add-on therapy based on physicians decision in accordance with summary of product characteristics (SmPC) and will be observed at baseline, 6 months (intermediate visit), and 12 months (final visit).
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets.
  Other Names: E2007; Fycompa
Drug: Perampanel — Perampanel oral suspension.
  Other Names: E2007; Fycompa

SUMMARY:
The primary purpose of this study is to investigate the effectiveness reflected by the retention rate of perampanel as the only add-on treatment in adult participants with primary generalized tonic-clonic (PGTC) or secondarily generalized tonic-clonic (SGTC) seizures based on focal or idiopathic generalized epilepsy in a non-interventional (observational) setting.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of epilepsy with PGTC or SGTC seizures based on focal or idiopathic generalized epilepsy
2. Active epilepsy with GTC seizures, demonstrated by the occurrence of at least 1 GTC seizure within 3 months before inclusion
3. The decision to prescribe perampanel was made by the physician before and irrespective of his/her decision to include the participant in the study
4. Receiving treatment with perampanel in line with the current Fycompa (perampanel) SmPC
5. Perampanel must either be newly administered as the only add-on treatment to a current antiepileptic drug (AED) monotherapy or must be planned to substitute one of two AEDs of a current dual therapy planned to be stopped within 2 months after initiation of treatment with perampanel. It will be specified which AED is planned to be substituted by perampanel upon inclusion. It is assumed that participants start treatment with perampanel closely after the baseline visit. Retrospective inclusions will be allowed, but only if the time between the initiation of perampanel treatment and inclusion does not exceed 7 calendar days. In this case, the baseline visit documentation should reflect the situation (including seizure situation 3 months before baseline and baseline medication) to the date perampanel treatment was initiated

Exclusion Criteria:

1. Participants with known psychogenic non-epileptic seizures
2. The participant had already received perampanel in the past
3. Simultaneous participation in an interventional clinical study and/or taking an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with PGTC or SGTC seizures.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Remaining on Perampanel at Month 12 (Retention Rate) | Month 12
  The retention rate is defined as the percentage of participants remaining on perampanel treatment at 12 months after the initiation of treatment.

SECONDARY OUTCOMES:
Percentage of Participants Remaining on Perampanel at Month 6 (Retention Rate) | Month 6
  The retention rate is defined as the percentage of participants remaining on perampanel treatment at 6 months after the initiation of treatment.
Percentage of Participants Who Achieved Seizure Freedom for All Generalized Tonic-clonic (GTC) Seizures at Month 12 | Month 12
Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Treatment-emergent Serious Adverse Events (SAE), and Adverse Events (AEs) by Severity | Up to Month 12
  AEs will be graded on a 3-point scale that is mild (discomfort noticed, but no disruption of normal daily activity), moderate (discomfort sufficient to reduce or affect normal daily activity), and severe (incapacitating, with inability to work or to perform normal daily activity).

CONTACTS AND LOCATIONS:
Locations (34):
- Germany (34):
  - Eisai Trial Site #51, Aalen
  - Eisai Trial Site #12, Berlin
  - Eisai Trial Site #43, Berlin
  - Eisai Trial Site #15, Bernau
  - Eisai Trial Site #8, Bielefeld
  - Eisai Trial Site #53, Bochum
  - Eisai Trial Site #38, Bonn
  - Eisai Trial Site #9, Bonn
  - Eisai Trial Site #25, Damp
  - Eisai Trial Site #48, Dortmund
  - Eisai Trial Site #27, Dresden
  - Eisai Trial Site #50, Dresden
  - Eisai Trial Site #7, Erlangen
  - Eisai Trial Site #44, Friedrichshafen
  - Eisai Trial Site #4, Greifswald
  - Eisai Trial Site #21, Hamburg
  - Eisai Trial Site #47, Hamburg
  - Eisai Trial Site #14, Jena
  - Eisai Trial Site #18, Kiel
  - Eisai Trial Site #54, Kiel
  - Eisai Trial Site #1, Kork
  - Eisai Trial Site #24, Leipzig
  - Eisai Trial Site #28, Lübeck
  - Eisai Trial Site #26, Magdeburg
  - Eisai Trial Site #13, Mainz
  - Eisai Trial Site #36, Mittweida
  - Eisai Trial Site #42, Nierstein
  - Eisai Trial Site #2, Radeberg
  - Eisai Trial Site #16, Ravensburg
  - Eisai Trial Site #23, Regensburg
  - Eisai Trial Site #46, Remscheid
  - Eisai Trial Site #3, Tübingen
  - Eisai Trial Site #37, Ulm
  - Eisai Trial Site #40, Weil der Stadt

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.